CLINICAL TRIAL: NCT01307033
Title: A Phase III, Randomized, Active-comparator Controlled and a Long-term Clinical Trial to Study the Safety of MK-0954A (L100/H12.5 mg) in Japanese Patients With Essential Hypertension Uncontrolled With MK-954H (L50/H12.5 mg) [PREMINENT®]
Brief Title: A Long-term Study of the Safety of MK-0954A in Patients With Essential Hypertension (MK-0954A-351)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-351
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Essential hypertension; Uncontrolled hypertension; Antihypertensive agents; Blood pressure
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-954H (L50/H12.5) (Active Comparator): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 50 mg (L50) and 12.5 mg of hydrochlorothiazide (H12.5). Participants will then receive open label MK-0954A (L100/H12.5) orally, once daily for 44 weeks (extension)
  Interventions: Drug: MK-954H; Drug: Placebo to MK-0954A
- MK-0954A (L100/H12.5) (Experimental): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 100 mg (L100) and 12.5 mg of hydrochlorothiazide (H12.5). Participants will continue to receive MK-0954A orally, once daily for 44 week extension
  Interventions: Drug: MK-0954A; Drug: Placebo to MK-954H

INTERVENTIONS:
Drug: MK-0954A — Tablet containing losartan potassium (100 mg) and hydrochlorothiazide (12.5 mg), once daily
  Arms: MK-0954A (L100/H12.5)
Drug: MK-954H — Tablet containing losartan potassium (50 mg) and hydrochlorothiazide (12.5 mg), once daily
  Other Names: Preminent®
  Arms: MK-954H (L50/H12.5)
Drug: Placebo to MK-0954A — Placebo tablet to match MK-0954A, once daily
  Arms: MK-954H (L50/H12.5)
Drug: Placebo to MK-954H — Placebo tablet to match MK-954H, once daily
  Arms: MK-0954A (L100/H12.5)

SUMMARY:
This study is being conducted to evaluate the safety of MK-0954A (L100/H12.5 mg) in essential hypertension participants who are uncontrolled with MK-954H (L50/H12.5 mg).

ELIGIBILITY:
Inclusion criteria:

* Participant has a diagnosis of essential hypertension.
* Participant is being treated with a single, or dual combination treatment for hypertension and will be able to discontinue the prior antihypertensive medication.
* Participant has a mean trough SiDBP of >=90mmHg and < 110mmHg.
* Participant has a mean trough SiSBP of >=140mmHg and < 200mmHg.
* Participant has no clinically significant abnormality at screening visit.

Exclusion criteria:

* Participant is currently taking > 2 antihypertensive medications.
* Participant has a history of significant multiple and/or severe allergies to ingredients of Nu-lotan or Preminent and thiazide drug or related drug (i.e., sulfonamide-containing "chlortalidone" medicines).
* Participant is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history within the last year of drug or alcohol abuse or dependence.
* Participant is pregnant or breastfeeding, or expecting to conceive or the pregnancy test is positive at screening visit.
* Participant is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-12-04 (Actual); Study Completion 2012-12-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rakugi H, Tsuchihashi T, Shimada K, Numaguchi H, Nishida C, Yamaguchi H, Fujimoto G, Azuma K, Shirakawa M, Hanson ME, Fujita KP. Efficacy and safety of losartan 100 mg/hydrochlorothiazide 12.5 mg in Japanese subjects with essential hypertension: two randomized, controlled trials. Hypertens Res. 2014 Dec;37(12):1042-9. doi: 10.1038/hr.2014.114. Epub 2014 Jul 3. PMID 24990091

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0954H (L50/H12.5) Double Blind Period (Period 1): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 50 mg (L50) and 12.5 mg of hydrochlorothiazide (H12.5)
- MK-0954A (L100/H12.5) Double Blind Period (Period 1): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 100 mg (L100) and 12.5 mg of hydrochlorothiazide (H12.5)
- L50/H12.5→L100/H12.5 Open Label (Period 2): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 50 mg (L50) and 12.5 mg of hydrochlorothiazide (H12.5). Participants will then receive open label MK-0954A (L100/H12.5) orally, once daily for 44 weeks (extension)
- L100/H12.5→L100/H12.5 Open Label (Period 2): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 100 mg (L100) and 12.5 mg of hydrochlorothiazide (H12.5). Participants will continue to receive MK-0954A orally, once daily for 44 week extension
Period: 8-week Double-blind Period
Arm/Group | MK-0954H (L50/H12.5) Double Blind Period (Period 1) | MK-0954A (L100/H12.5) Double Blind Period (Period 1) | L50/H12.5→L100/H12.5 Open Label (Period 2) | L100/H12.5→L100/H12.5 Open Label (Period 2)
Started | 144 | 134 | 0 | 0
Completed | 131 | 127 | 0 | 0
Not Completed | 13 | 7 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Blood Pressure Withdrawal Criteria Met | 0 | 3 | 0 | 0
Not completed — Potassium Withdrawal Criteria Met | 6 | 3 | 0 | 0
Period: 44-week Open-label Extension
Arm/Group | MK-0954H (L50/H12.5) Double Blind Period (Period 1) | MK-0954A (L100/H12.5) Double Blind Period (Period 1) | L50/H12.5→L100/H12.5 Open Label (Period 2) | L100/H12.5→L100/H12.5 Open Label (Period 2)
Started | 0 | 0 | 131 | 127
Completed | 0 | 0 | 120 | 115
Not Completed | 0 | 0 | 11 | 12
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Blood Pressure Withdrawal Criteria Met | 0 | 0 | 0 | 2
Not completed — Potassium Withdrawal Criteria Met | 0 | 0 | 6 | 7
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-0954H (L50/H12.5): One combination tablet daily, orally, for 8 weeks. Each tablet contains Losartan 50 mg (L50) and 12.5 mg of hydrochlorothiazide (H12.5). Participants will then receive open label MK-0954A (L100/H12.5) orally, once daily for 44 weeks (extension)
- Total: Total of all reporting groups
Arm/Group | MK-0954H (L50/H12.5) | MK-0954A (L100/H12.5) | Total
Number analyzed (Participants) | 144 | 134 | 278
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (10.7) | 57.8 (10.8) | 57.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 32 | 73
  Male | 103 | 102 | 205

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 8
Description: Blood pressure (BP) was measured with an automatic sphygmomanometer after participant has been resting in a sitting position for at least 10 minutes. BP was determined averaging 3 replicate measurements obtained at least a 1- to 2-minute interval between BP measurements. The recorded BP was the calculated average of the 3 readings.
Time Frame: Baseline and Week 8 (End of Double-blind Period)
Population: Full Analysis Set (FAS) population: defined as all randomized participants who received at least one dose of study treatment, had at least one post-randomization observation for the analysis endpoint subsequent to at least one dose of study treatment, and had baseline data for those analyses that required baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- MK-0954H (L50/H12.5): One combination tablet daily for 8 weeks. Each tablet contains Losartan 50 mg (L50) and 12.5 mg of hydrochlorothiazide (H12.5).
- MK-0954A (L100/H12.5): One combination tablet daily for 8 weeks. Each tablet contains Losartan 100 mg (L100) and 12.5 mg of hydrochlorothiazide (H12.5).
Arm/Group | MK-0954H (L50/H12.5) | MK-0954A (L100/H12.5)
Number analyzed (Participants) | 144 | 134
mmHg | -5.3 (0.7) [-6.6 to -3.9] | -5.0 (0.7) [-6.4 to -3.6]
Statistical Analysis 1: Comparison: MK-0954H (L50/H12.5) vs MK-0954A (L100/H12.5); Test type: Superiority or Other; Constained logitudinal data analysis; Model included treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups; Difference in least squares means = 0.2, 95% CI 2-sided [-1.7 to 2.2]

2. Secondary Outcome: Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) at Week 8
Description: as for outcome 1
Time Frame: Baseline and Week 8 (End of Double-blind Period)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-0954H (L50/H12.5) | MK-0954A (L100/H12.5)
Number analyzed (Participants) | 144 | 134
mmHg | -6.2 [-8.2 to -4.3] | -8.5 [-10.5 to -6.5]
Statistical Analysis 1: Comparison: MK-0954H (L50/H12.5) vs MK-0954A (L100/H12.5); Test type: Superiority or Other; Constained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.3, 95% CI 2-sided [-5.0 to 0.5]

3. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event When Receiving MK-0954A (L100/H12.5) During Study (8-week Double-blind and/or 44-week Open-label Extension)
Time Frame: Up to 52 weeks
Population: All-Patients-as-Treated (APaT) Population, which consists of all randomized patients who received at least one dose of MK-0954A. The L100/H12.5 (L50/H12.5) arm only includes data from extension period (44 weeks); L100/H12.5→L100/H12.5 Open Label arm includes data from entire study period (52 weeks).
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5→L100/H12.5 Open Label (Period 2) | L100/H12.5→L100/H12.5 Open Label (Period 2)
Number analyzed (Participants) | 131 | 134
Percentage of Participants | 71.0 | 72.4

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: All-Patients-as-Treated (APaT) Population defined as all randomized participants who received at least one dose of study treatment.
Arm/Group | MK-0954H (L50/H12.5) Double Blind Period (Period 1) | MK-0954A (L100/H12.5) Double Blind Period (Period 1) | L50/H12.5→L100/H12.5 Open Label (Period 2) | L100/H12.5→L100/H12.5 Open Label (Period 2)
Serious Adverse Events (participants affected / at risk) | 1/144 | 2/134 | 6/131 | 1/127
Other Adverse Events (participants affected / at risk) | 18/144 | 20/134 | 47/131 | 43/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0954H (L50/H12.5) Double Blind Period (Period 1) (N=144) | MK-0954A (L100/H12.5) Double Blind Period (Period 1) (N=134) | L50/H12.5→L100/H12.5 Open Label (Period 2) (N=131) | L100/H12.5→L100/H12.5 Open Label (Period 2) (N=127)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0954H (L50/H12.5) Double Blind Period (Period 1) (N=144) | MK-0954A (L100/H12.5) Double Blind Period (Period 1) (N=134) | L50/H12.5→L100/H12.5 Open Label (Period 2) (N=131) | L100/H12.5→L100/H12.5 Open Label (Period 2) (N=127)
Nasopharyngitis (Infections and infestations) | 11 (13) | 10 (11) | 22 (36) | 27 (34)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 10 (10) | 7 (7)
Blood uric acid increased (Investigations) | 7 (7) | 8 (8) | 6 (6) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7) | 5 (5)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 7 (8) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.